CLINICAL TRIAL: NCT00555932
Title: Utility of Modern Ultrasound Techniques in the Evaluation of Cerebral Venous Sinuses in Neonates
Brief Title: Modern Ultrasound Techniques in the Evaluation of Cerebral Venous Sinuses in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Manohar Shroff, Chief, Diagnostic Imaging, Pediatric Neuroradiologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1000010745
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Intracranial Thrombosis
Keywords: Intracranial Thrombosis; Cerebral Sinovenous Thrombosis; Pediatrics; Cranial Ultrasound
MeSH Terms: conditions — Intracranial Thrombosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): The research head ultrasound (HUS) will be performed at the bedside in the Neonatal Unit. The ultrasound examination will be performed within 10 hours time window of the MR and or CT study.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — All the studies will be performed with the portable ultrasound machine used on a regular basis in the neonatal care unit.

SUMMARY:
Our overall aim is to examine if ultrasound is as accurate as MRI and/or CT in the evaluation of dural venous sinuses. We hypothesize that sonography will be accurate (accuracy >80%) for diagnosing specific anatomic findings of dural venous sinuses.

DETAILED DESCRIPTION:
Cranial ultrasound is an established technique for evaluation of the neonatal brain. However its role in the evaluation of cerebral dural venous sinuses in neonates has not been established. It is very important to evaluate the cerebral dural venous sinuses, as cerebral sinovenous thrombosis (CSVT) is an increasingly recognized condition in neonates.

There is an obvious clinical need for systematically evaluating the role of ultrasound with doppler in the evaluation of cerebral venous sinuses. Advances in diagnostic imaging have led to rapid clinical implementation of newer technologies like MR and CT for evaluation of venous sinuses. However technological advances in older imaging methods like ultrasound which have advantages of being non-invasive and being performed at the bedside have not been evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. All neonates (up to 28 days old) and preterm infants, hospitalized at HSC who need clinically indicated brain MR and MRV as part of their diagnostic workup. Clinical indications for MR could include birth asphyxia, seizures, irritability, lethargy, abnormal neurological examination, etc.
2. Neonates and preterm infants & who are clinically considered stable to undergo the ultrasound study. This will be determined at the bedside by the neonatology team in attendance.
3. Where consent is available from parents.
4. Only neonates and preterm infants who have undergone a technically adequate MRI study which includes vascular MR venography sequences or CT with contrast will be included. Assessments for technically adequacy will be made by the technologist or the supervising radiologist, as per clinical protocols currently used in the department of diagnostic imaging. This will be determined by referring to notes made on the request form and also by direct communication between the supervising radiologist and team members obtaining consent.

Exclusion Criteria:

1. Vital signs will be monitored in the usual manner by the nurses in attendance in the neonatal unit. If the neonate is unstable, an ultrasound study will not be done.
2. If after starting the ultrasound, any signs of instability are noted during the study, the ultrasound study will discontinued.
3. If consent from parent or guardian is not available, the research ultrasound study will not be done.
4. If the ultrasound cannot be done within a 10 hours window of the CT or MR study (due to technical problems with machine or skilled personnel not being available).
5. Neonates & preterm infants who have undergone technically inadequate MR and/or CT will not be included. Such technical inadequacy will be determined by referring to notes made by the technologist on the request form and by direct communication with the supervising radiologist.
6. Neonates & preterm infants undergoing repeat CT and/or MRs will be excluded from the study.

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To prospectively evaluate the feasibility of visualization of normal dural venous sinuses, their patency, and normal variations with ultrasound in newborn children (preterm & term), using cross sectional imaging (MRI and/or CT) as reference standards. | Within 10 hours of the MRI scan

SECONDARY OUTCOMES:
The ability of doppler ultrasound to evaluate flow velocities in all dural venous sinuses that will be evaluated in this study. | Within 10 hours of MRI

CONTACTS AND LOCATIONS:
Overall Officials: Manohar Shroff, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Link to final publication abstract — http://www.ncbi.nlm.nih.gov/pubmed/22532234